CLINICAL TRIAL: NCT06652659
Title: Risk Factors for Development of Non-union of Displaced Midshaft Clavicle Fractures: A Prospective Double-center Cohort Study
Brief Title: Risk Factors for Development of Non-union of Displaced Midshaft Clavicle Fractures
Acronym: RisC
Status: Recruiting | Type: Observational
Sponsor: Bispebjerg Hospital (Other)
Responsible Party: Principal Investigator, Ida Tryggedsson, Medical doctor, principal investigator, Bispebjerg Hospital
Other Study IDs: H-24022926
Record Dates: First submitted 2024-10-18; First posted 2024-10-22 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-02

CONDITIONS: Non-union of Fractures
Keywords: Non-union; Midshaft Clavicle Fracture; Clavicle; Midshaft; Midshaft Clavicle; Risc Factors for Non-union

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Biospecimen Retention: Samples Without DNA — General health biomarkers. Bone health biomarkers.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients at age 18 or above with a displaced midshaft clavicle fracture.
  Interventions: Other: Non-union

INTERVENTIONS:
Other: Non-union — Observational study looking prospectively at many different factors that may affect non-union of midshaft clavicle fractures.

SUMMARY:
Clavicle fractures are common and usually heal well without surgery. Most patients recover full shoulder function within a few weeks with conservative treatment, which is the standard in Denmark. However, in cases where the broken ends of the bone do not touch (displaced fractures), there is a higher risk of complications like non-healing (non-union), affecting 11-18% of such cases. Non-union can lead to long-term pain, reduced shoulder function, and a longer recovery time, often requiring multiple follow-up visits.

While surgery might prevent these complications for some patients, operating on all displaced fractures would lead to overtreatment. The current challenge is identifying which patients are at risk for non-union and would benefit most from surgery. This study aims to investigate the risk factors for non-union in patients with displaced clavicle fractures by examining both patient characteristics and fracture-related factors.

The goal is to use multiple data points to develop a score that can support clinicians and patients in shared decision-making regarding the optimal and individualized treatment for clavicle fractures.

This research is important not only for clavicle fractures but also for understanding and treating non-union in other bones like the ulna and tibia, which face similar challenges.

DETAILED DESCRIPTION:
Clavicle fracture The clavicle, the collarbone, connects the arm to the axial skeleton. It is essential to shoulder function as it provides attachment for the primary muscles stabilizing the shoulder joint, and allows an extensive range of motion by the upper limb.

The clavicle fracture is a common skeletal injury that accounts for approximately 5% of all adult fractures and 35-40% of injuries to the shoulder girdle. According to extensive epidemiological studies, the majority of clavicle fractures occur in the middle third, with 50-70% of those being displaced. It means that for every 100 clavicle fractures, approximately half of them are displaced midshaft fractures.

A clavicle fracture is frequently caused by a direct impact to the shoulder, often resulting from same-level falls, bicycle accidents, or sports-related incidents, which makes it a common fracture in Denmark. There is a classic bimodal distribution of the fracture with increased incidence in younger males, usually due to high-energy trauma, and a second peak in the elderly population often associated with low-energy falls. According to the Danish Health Data Authority, the incidence of clavicle fractures is relatively high, approximately 65/100,000 from 1996-2018, and numbers have been increasing throughout the years.

Most clavicle fractures heal uneventfully and are traditionally treated non-operatively with immobilization in an arm sling for a few weeks, typically attaining full recovery and range of motion within six weeks.

Clavicle non-union Fracture non-union is a rare but severe complication that affects 5-10% of all fractures worldwide, depending on fracture location and country. The risk of non-union is higher when the fracture is displaced and bone ends shift out of their normal alignment, especially in the clavicle, which has one of the highest rates of non-union. Non-union can cause long-term pain, physical disability, reduced quality of life, and an extended recovery period before returning to regular work productivity. Often a non-union requires later complex operative treatment.

Although the incidence of non-union in the clavicle is approximately 10%, performing surgery on all displaced clavicle fractures would lead to overtreatment of fractures that would have healed uneventfully without surgery. Therefore, it is essential to identify patients predisposed to non-union and the risk factors involved to personalize the initial treatment. However, it is a major clinical challenge to identify these patients.

Recent studies on clavicle fractures have focused on comparing the outcomes of non-operative and operative treatment. Despite various randomized controlled trials, a Cochrane review from 2019 concluded that there is limited evidence for choosing one treatment over the other and that the choice of care must be determined on an individual patient basis.

Risk factors Various studies have examined the predictors associated with non-union, and many have found it to be a multifactorial issue. The degree of displacement, or the distance between bone ends, is usually the most significant factor in predicting non-union. Other risk factors include female gender, older age, smoking, persistent pain, fracture comminution, fracture shortening, and absence of developing bridging callus at the fracture site. Typically, the more risk factors present, the greater the risk of non-union. When evaluating patient-related factors, studies usually look at factors related to the host's physiological state, including gender, age, comorbidities, smoking and alcohol status, weight, BMI, and occupation. To cover patient-related factors, it is also necessary to assess the patient's molecular environment, meaning biomarkers for bone health to be found in the blood.

Rationale Research exploring risk factors that predispose patients to the development of symptomatic non-union of clavicle fractures is lacking. Before treatment can be individualized, clinical studies assessing possible risk factors are needed to fill this knowledge gap.

Hypothesis Patients suffering a displaced midshaft clavicle fracture are not at equal risk of development of non-union following conservative treatment.

10% is expected to develop a non-union within 6 months following the injury and the investigators expect to uncover specific clinical, radiological and molecular risk factors for non-union.

Purpose

Overall aim:

The purpose of this study is to identify risk factors for the development of non-union following a displaced midshaft clavicle fracture. The investigators aim to combine clinical, radiological, and molecular risk factors for the establishment of a predictive risk score that may help to assess individual susceptibility to non-union. A risk score combining all aspects will be a practical tool to aid clinicians in identifying and managing patients with increased risk of non-union at the time of initial presentation. This enables individualized treatment and a chance to improve overall outcome for the patient.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age upon study enrollment
* Admitted to the emergency room (ER) at BBH or HVH with a displaced midshaft clavicle fracture
* Danish social security number
* Understand Danish
* Able to fill out questionnaire by hand or online.
* Provides informed consent prior to initiation of any study-related activities/procedures

Exclusion Criteria:

* Subject incapable of understanding the patient information or unable to provide informed consent
* Open fracture or fracture with risk of skin penetration
* Pathological fracture
* Clavicle fracture due to polytrauma
* Floating shoulder injury
* Vascular injury at fracture site
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients at age 18 years or above with a displaced midshaft clavicle fracture in the are of Bispebjerg Hospital and Hvidovre Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2024-10-21 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Radiographic Non-Union assessed by 2-plane radiograph at 26 weeks post-injury | 26 weeks
  Measure: Radiographic assessment of non-union using standard 2-plane radiographs at 26 weeks post-injury.
  Non-Union Assessment: Non-union will be defined as the absence of bridging callus on radiographs at 6 months post-injury, measured on standard 2-plane radiographs of the clavicle. The assessment will include measurement of displacement and shortening (measured in millimeters).

SECONDARY OUTCOMES:
Visual Analog Scale (VAS) score | Week 1 to week 6
  Measure: The Visual Analog Scale (VAS) score is used to measure a person's subjective experience of pain on a scale from 0 to 10, with 0 being no pain and 10 being the worst possible pain. Participants will record a VAS-score daily from week 1 to week 6.
  Purpose: To investigate if patients who suffer prolonged pain and thus will not show a significant improvement in Visual Analog Scale (VAS) score within 6 weeks from injury are predisposed to the development of non-union.
Shoulder function measured by the quick Disabilities of the Arm, Shoulder and Hand (qDASH) score | 1 week, 6 weeks, 12 weeks, 26 weeks, 52 weeks
  Measure: The quick Disabilities of Arm Shoulder Hand (qDASH) measures physical function and symptoms in people with musculoskeletal disorders of the upper limb. The qDASH consists of 11 items that patients rate on a scale of 1 (no difficulty or no symptoms) to 5 (extreme difficulty or severe symptoms). The responses are averaged and then transformed into a score on a scale from 0 to 100.
  Purpose: To investigate if patients who do not show a significant improvement in range of motion of the shoulder and no significant increase in qDASH score are predisposed to development of non-union.
Quality of Life measured by the EuroQol (EQ-5D-5L) questionnaire | 1 week, 6 weeks, 12 weeks, 26 weeks, 52 weeks.
  Measure: The EuroQol (EQ-5D-5L) questionnaire is used to assess patient-reported outcomes related to health-related quality of life. It evaluates five dimensions, each rated on a 5-point scale, where 1 represents no issues and 5 represents severe issues. The EQ-5D-5L can describe up to 3,125 different health states. A score of 11111 signifies no problems in any dimension, while a score of 55555 reflects extreme problems across all dimensions.
  Purpose: To investigate whether patients who do not show significant improvement in their EQ-5D-5L score are at increased risk of developing non-union following non-operative treatment.
Radiographic assessment of fracture characteristics | 1 week, 6 weeks, 12 weeks, 26 weeks, 52 weeks
  Measure: Radiographic assessment of non-union using standard 2-plane radiographs. Assessment will include description of callus formation (binary: yes/no) and measurement of displacement and shortening (millimeter).
Plasma concentration of health-related biomarkers | 1 week
  Measure: Blood sample collected at 1 week post injury. The sample will be analyzed for concentration of 25-hydroxyvitamin D, Calcium, Phosphorus, Bone-specific Alkaline Phosphatase, Alkaline Phosphatase, Magnesium, HbA1c, Intact parathyroid hormone, Insulin-like growth factor 1, Thyroid function tests, Free testosterone, Estradiol, Complete blood count (CBC), P1NP (procollagen), osteocalcin, calcitonin, CGRP, RAKL, sclerostin.
  Purpose: To assess if any abnormal levels of biomarkers at 1 week affect development of non-union at 26 weeks.
Patient-related factors extracted from medical record | Week 1
  Measure: Data extracted from patient medical records including demographic information, gender, height, weight, smoking status, weekly alcohol consumption, medicine use, comorbidities, and employment status Purpose: To investigate if any patient-related factors present at week 1 predispose for development of non-union at 26 weeks.

CONTACTS AND LOCATIONS:
Locations (2):
- Denmark (2):
  - Bispebjerg Hospital, Copenhagen NV
  - Hvidovre Hospital, Hvidovre

IPD SHARING:
Plan to Share IPD: No
Not allowed due to study approval from national ethics comite.

REFERENCES:
- [Background] Qvist AH, Vaesel MT, Jensen CM, Jakobsen T, Jensen SL. Minimal Pain Decrease Between 2 and 4 Weeks After Nonoperative Management of a Displaced Midshaft Clavicle Fracture Is Associated with a High Risk of Symptomatic Nonunion. Clin Orthop Relat Res. 2021 Jan 1;479(1):129-138. doi: 10.1097/CORR.0000000000001411. PMID 32675585
- [Background] Ban I, Troelsen A. Risk profile of patients developing nonunion of the clavicle and outcome of treatment--analysis of fifty five nonunions in seven hundred and twenty nine consecutive fractures. Int Orthop. 2016 Mar;40(3):587-93. doi: 10.1007/s00264-016-3120-8. Epub 2016 Feb 4. PMID 26847264
- [Background] Nicholson JA, Oliver WM, MacGillivray TJ, Robinson CM, Simpson AHRW. Sonographic bridging callus at six weeks following displaced midshaft clavicle fracture can accurately predict healing. Bone Joint Res. 2021 Feb;10(2):113-121. doi: 10.1302/2046-3758.102.BJR-2020-0341.R1. PMID 33543996
- [Background] Liu W, Xiao J, Ji F, Xie Y, Hao Y. Intrinsic and extrinsic risk factors for nonunion after nonoperative treatment of midshaft clavicle fractures. Orthop Traumatol Surg Res. 2015 Apr;101(2):197-200. doi: 10.1016/j.otsr.2014.11.018. Epub 2015 Feb 18. PMID 25703151
- [Background] Jorgensen A, Troelsen A, Ban I. Predictors associated with nonunion and symptomatic malunion following non-operative treatment of displaced midshaft clavicle fractures--a systematic review of the literature. Int Orthop. 2014 Dec;38(12):2543-9. doi: 10.1007/s00264-014-2450-7. Epub 2014 Jul 16. PMID 25027978
- [Background] Lenza M, Buchbinder R, Johnston RV, Ferrari BA, Faloppa F. Surgical versus conservative interventions for treating fractures of the middle third of the clavicle. Cochrane Database Syst Rev. 2019 Jan 22;1(1):CD009363. doi: 10.1002/14651858.CD009363.pub3. PMID 30666620
- [Background] Axelrod DE, Ekhtiari S, Bozzo A, Bhandari M, Johal H. What Is the Best Evidence for Management of Displaced Midshaft Clavicle Fractures? A Systematic Review and Network Meta-analysis of 22 Randomized Controlled Trials. Clin Orthop Relat Res. 2020 Feb;478(2):392-402. doi: 10.1097/CORR.0000000000000986. PMID 31574019
- [Background] Zura R, Xiong Z, Einhorn T, Watson JT, Ostrum RF, Prayson MJ, Della Rocca GJ, Mehta S, McKinley T, Wang Z, Steen RG. Epidemiology of Fracture Nonunion in 18 Human Bones. JAMA Surg. 2016 Nov 16;151(11):e162775. doi: 10.1001/jamasurg.2016.2775. Epub 2016 Nov 16. PMID 27603155
- [Background] Yan MZ, Yuen WS, Yeung SC, Wing-Yin CW, Wong SC, Si-Qi WW, Tian E, Rashed S, Yung CSY, Fang CX. Operative management of midshaft clavicle fractures demonstrates better long-term outcomes: A systematic review and meta-analysis of randomised controlled trials. PLoS One. 2022 Apr 29;17(4):e0267861. doi: 10.1371/journal.pone.0267861. eCollection 2022. PMID 35486618
- [Background] Ban I, Branner U, Holck K, Krasheninnikoff M, Troelsen A. Clavicle fractures may be conservatively treated with acceptable results - a systematic review. Dan Med J. 2012 Jul;59(7):A4457. PMID 22759840
- [Background] Hill JM, McGuire MH, Crosby LA. Closed treatment of displaced middle-third fractures of the clavicle gives poor results. J Bone Joint Surg Br. 1997 Jul;79(4):537-9. doi: 10.1302/0301-620x.79b4.7529. PMID 9250733
- [Background] Nowak J, Mallmin H, Larsson S. The aetiology and epidemiology of clavicular fractures. A prospective study during a two-year period in Uppsala, Sweden. Injury. 2000 Jun;31(5):353-8. doi: 10.1016/s0020-1383(99)00312-5. PMID 10775691
- [Background] Moverley R, Little N, Gulihar A, Singh B. Current concepts in the management of clavicle fractures. J Clin Orthop Trauma. 2020 Feb;11(Suppl 1):S25-S30. doi: 10.1016/j.jcot.2019.07.016. Epub 2019 Jul 24. PMID 31992912